CLINICAL TRIAL: NCT05995613
Title: Evaluation of Wearable Melanin-Adjusted Blood Oxygen Sensor (MABOS) for Improved Accuracy in Patients of Color
Brief Title: Evaluation of MABOS for Improved Pulse Oximeter Accuracy in Patients of Color
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 23-0812
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2023-08

CONDITIONS: Oxygen Saturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MABOS: Participants will have one FDA-approved pulse oximeter (Nonin PureSat) along with our novel pulse oximeter placed to acquire 90 minutes of biometric data
  Interventions: Device: MABOS; Device: Nonin PureSat

INTERVENTIONS:
Device: MABOS — The novel pulse oximeter (MABOS) will be placed to acquire two biometrics: blood oxygen saturation and epidermal melanin concentration.
  Other Names: pulse oximeter
Device: Nonin PureSat — An FDA approved pulse oximeter will be placed to acquire blood oxygen saturation.

SUMMARY:
Purpose: Investigate the safe wearability and basic functionality - epidermal melanin concentration and blood oxygen estimation - of our developed device: Melanin-Adjusted Blood Oxygen Sensor (MABOS)

Participants: Healthy adults 18-65 years of age

Procedures (methods): The investigators plan to enroll 12 healthy adult participants for the study. The investigators aim to enroll 4 participants with skin tones associated with those of African descent (Group A), 4 of East Asian descent (Group B), and 4 of European descent (Group C). Additionally, the investigators aim to ensure half of group is male, and the other half female. For the duration of the study, two wearable devices will be placed on the participant: a Nonin PureSat pulse oximeter on a forefinger, and the novel wearable pulse oximeter - MABOS - on the other forefinger. Prior to testing, an Ocean HR2 XR Spectrometer will be used to assess the absorbance of three wavelengths of light - 410, 660, 940 nm - on each patient's inner wrist. Following this, the two devices will be placed on the patient, set up, and calibrated for 10 minutes. During the calibration period, MABOS will be used to measure the same three wavelengths of light utilized by the Ocean HR2 XR Spectrometer (410, 660, and 940 nm). After the calibration period, all participants will be asked to perform the following procedure 5 times as part of the testing period: a deep inhalation lasting no longer than 10 seconds, followed by a slow exhalation lasting no longer than 30 seconds. Between each trial, a five-minute break will be required. For the entire testing period, all two devices will be continuously acquiring data. After this testing period, all two devices will continue taking measurements until 90 minutes have elapsed. Skin integrity will be examined before spectrometer use, after spectrometer use, after the calibration period, every 30 minutes after the start of the testing period, and after the testing period. During the study, if the participants report any uncomfortable feeling and/or pain or if a change to the skin at the site of device placement occurs, the measurements will be discontinued, and all the devices placed on the participants will be removed. Questionnaires will be provided after the study period and during follow-up visits approximately 48 hours and 96 hours post the device testing visit for a proof-of-concept evaluation of the safe wearability.

ELIGIBILITY:
Inclusion Criteria:

* Male and females, with age between 18-65
* Health individuals (defined as: not known to suffer any significant illnesses relevant to the proposed study, cited from The Textbook of Pharmaceutical Medicine)
* The investigators aim to enroll 4 participants with skin tones associated with those of African descent, 4 of East Asian Descent, and 4 of European Descent. Additionally, the investigators aim to ensure half of the group is male, the other half female.

Exclusion Criteria:

* Pregnant or lactating
* History of active (clinically significant) skin disorders that make skin vulnerable to contact conventional electronic devices.
* History of allergic response to silicones or adhesives (such as 3M Tegaderm)
* Broken, damaged, or irritated skin or rashes near the sensor application sites
* Subjects who are physically or cognitively unable to perform activities of daily living, assessed at the discretion of the investigator to ensure safe completion of study tasks.
* Inability to perform the breathing tests - deep inhalation for 10 seconds, followed by a slow exhalation no longer than 30 seconds.
* Presence of tattoos on fingers, hands, or forearms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals of African, East Asian, and European descent; equal proportions of male and female individuals from each group.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Initial Device Safety Questionnaire | 10 minutes following the 90 minute testing period
  Device safety and comfort will be assessed by qualitative survey. All questions are rated from 1-5, where 1 is Strongly Disagree, and 5 is Strongly Agree. In the initial survey, the final 7 pertain to safety.
  The Safety Sub-Score is determined by the latter 7 questions, making the score range from 7-35.
  In this case, a higher number indicates a better outcome.
Initial Device Comfort Questionnaire | 10 minutes following the 90 minute testing period
  Device comfort will be assessed by qualitative survey. All questions are rated from 1-5, where 1 is Strongly Disagree, and 5 is Strongly Agree. In the initial 19-question survey, the first 12 pertain to comfort.
  The Comfort Sub-Score is determined by the first 12 questions, making the score range from 12-60.
  In this case, a higher number indicates a better outcome.
Final Device Safety Questionnaire | Two 10-minute sessions, one 2 days after the testing session, and one 4 days after the testing session
  Device safety will be assessed by qualitative survey. All questions are rated from 1-5, where 1 is "Strongly Disagree", and 5 is "Strongly Agree" and scores range from 9-45, where a higher score indicates a better outcome. The following 9 questions are asked: "I have noticed a change in skin condition since wearing the device"; "I have experienced a rash since wearing the device"; "I have experienced itching since wearing the device"; "I have experienced swelling since wearing the device"; "I have experienced a burning sensation since wearing the device"; "I have experienced vesicles blistering since wearing the device"; "I have experienced irregular warming of the skin since wearing the device"; "I have experienced a stinging sensation since wearing the device"; and "I have experienced a change in skin sensitivity since wearing the device."

SECONDARY OUTCOMES:
Epidermal Melanin Estimation | First 10 minutes of the 90-minute testing session, during the calibration phase
  Confirming the device's ability to differentiate skin tone using 3 wavelengths of light by comparison to a spectrometer.
  Metric of Accuracy: Take the average 410 nm light absorption of each individual (an average of intensity of absorbance over time during the 10-minute calibration period), using both the spectrometer and the device. Find the regression line that best fits the 12 data points (where each data point is a paired observation of spectrometer and device 410-nm light absorption for a given participant). A positive R value, with an R-squared value >80% for a simple linear regression, is considered a positive indication of a trend.
Blood Oxygen Level Estimation | The latter 80 minutes of the testing period on the testing day, following the calibration period
  Comparing the device's blood oxygen estimation to the FDA approved device to confirm accuracy.
  Metric of Accuracy: Upon calibration of the device, each 60-second sample will constitute one 'estimate' of SpO2 (blood oxygen saturation). For the latter 80 minutes of the study, 80 samples will be derived. Each sample will be compared to what was recorded by the FDA-approved oximeter. The comparison will be accomplished by finding the regression line that best fits the cumulative 80-minute data from all 12 participants. A positive R value, with an R-squared value >80% for a simple linear regression, is considered a positive indication of a trend.

CONTACTS AND LOCATIONS:
Overall Officials: Wubin Bai, Ph.D., Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No